CLINICAL TRIAL: NCT03944252
Title: Randomized Phase 2 Trial of Cetuximab and Avelumab or Avelumab Alone for Unresectable, Locally Advanced or Metastatic Squamous Cell Anal Carcinoma (SCCAC) Progressed After at Least One Line of Systemic Treatment
Brief Title: Cetuximab + Avelumab or Avelumab Alone for Unresectable, Locally Advanced or Metastatic Squamous Cell Anal Carcinoma (SCCAC) Progressed After at Least One Line of Systemic Treatment (CARACAS)
Acronym: CARACAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-000737-12
Record Dates: First submitted 2019-04-12; First posted 2019-05-09 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Squamous Cell Anal Carcinoma
MeSH Terms: conditions — Anus Neoplasms | interventions — avelumab; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (avelumab) (Experimental): avelumab 10 mg/kg iv day 1; To be repeated every 2 weeks (14 days) until progression of disease, refuse or inacceptable toxicity.
  Interventions: Drug: Avelumab
- B (cetuximab + avelumab) (Experimental): cetuximab 500 mg/m2 plus avelumab 10 mg/kg iv day 1. To be repeated every 2 weeks (14 days) until progression of disease, refuse or inacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Avelumab — avelumab 10 mg/kg iv day 1; To be repeated every 2 weeks (14 days) until progression of disease, refuse or inacceptable toxicity.
Drug: Cetuximab — cetuximab 500 mg/m2 plus avelumab 10 mg/kg iv day 1. To be repeated every 2 weeks (14 days) until progression of disease, refuse or inacceptable toxicity.
  Arms: B (cetuximab + avelumab)

SUMMARY:
* The standard first line treatment in SCCAC is the association of 5-FU with cisplatin reaching a percentage of survival at 5 years of about 32% (Faivre 1999); in a recent case series of patients affected by SCCAC, the combination of 5-FU and cisplatin as first line treatment produced 34.4% objective response rate (ORR) and a 5 years survival rate of 15% (Sclafani 2017);
* No standard second line treatment exists for SCCAC;
* Cetuximab in association with irinotecan has demonstrated promising results in pretreated patients affected by SCCAC (Lukan 2009). In addition, it was recently tested in stage I-III SCCAC in association with cisplatin plus 5-FU and radiotherapy. Despite not reaching their pre-specified endpoints both studies reported an interesting activity in local control of disease, leading to hypothesize that cetuximab warrant further investigation in new strategies (Garg 2017, Sparano 2017);
* Anti-PD1 treatments such as nivolumab and pembrolizumab showed promising activity in metastatic refractory SCCAC in terms of response rate and disease control with acceptable toxicity profiles (Morris 2017, Ott 2017);
* The induction of immunogenic cell death was recently shown for cetuximab-based regimens (Pozzi 2016) and PD-L1 blockade should lead to NK cells activation enhancing cetuximab ADCC (Concha-Benavente 2015, Concha-Benavente 2016).

On the basis of these considerations, the investigators designed the present randomized phase II trial of avelumab alone or avelumab plus cetuximab for previously treated unresectable locally advanced or metastatic SCCAC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of SCCAC;
* Progression on or after first line systemic therapy for surgically unresectable or metastatic disease. Systemic radiosensitizing chemotherapy with curative intent in limited-stage disease should be considered equal to a first line for a patient experiencing progression during or within 6 months of completion;
* Evaluable disease lesion according to RECIST v1.1 criteria;
* Availability of tumor sample (primary and/or metastatic sites);
* Age ≥ 18 years;
* Eastern Cooperative Oncology Group - Performance Status (ECOG PS) ≤ 2;
* Life expectancy of at least 12 weeks;
* Laboratory Requirements:

Neutrophils ≥ 1.5 x 109 /L; Platelets ≥ 100 x 109 /L; Hemoglobin ≥ 9 g/dL; Total bilirubin ≤ 1.5 time the upper-normal limits (UNL) of the normal values and ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases); Alkaline phosphatase ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases); Creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) or serum creatinine ≤1.5 x UNL;

* HIV-positive patients are eligible if their CD4+ cell count amounts to 300 cells per μL or more; HIV viral load has to be undetectable, and they have to be compliant with antiretroviral treatment;
* Negative serum or urine pregnancy test at screening for women of childbearing potential. Female subjects, or male subjects with female partners of child-bearing potential must be willing to use highly effective contraception as approved by the investigator (i.e. barrier contraceptive measure or oral contraception, total abstinence) during the study and until 30 days after last study treatment;
* Written informed consent to the study procedures and to molecular analyses before patients registration;
* Will and ability to comply with the protocol.

Exclusion Criteria:

* Previous therapy with any drug targeting T-cell co-regulatory proteins (i.e., immune checkpoint inhibitors);
* Concurrent anticancer treatment or use of any investigational drug within 28 days before the start of the trial treatment;
* Major surgical procedure, open biopsy, or significant traumatic injury occurred within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study;
* History or evidence upon physical examination of CNS disease unless adequately treated. Patients with treated brain metastases are eligible if their lesions were stable and asymptomatic for at least 3 months;
* Neutrophils < 1.5 x 109/L; Platelets < 100 x 109/L; Hemoglobin < 9 g/dL;
* Active uncontrolled infections requiring systemic therapy or other clinically relevant concomitant illness contraindicating therapy administration or putting the patient at high risk for treatment-related toxicities;
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive);
* Patients with active autoimmune disease or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent or might potentially affect vital organ function, or require use of immunosuppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use for ≥ 1 month). Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible;
* Current use of immunosuppressive medication, EXCEPT for the following:

  1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication);
* Prior organ transplantation including allogenic stem-cell transplantation;
* Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines;
* Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma;
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication;
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonia, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable;
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma of the skin or cervical cancer in situ;
* Pregnant or lactating women;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is Objective Response Rate (ORR). | Radiological responses will be evaluated starting from cycle 1 day 1 of treatment until disease progression, withdrawal of consent or death for any reason, whichever occurs first assessed up to 12 moths.
  The primary endpoint is Objective Response Rate (ORR). ORR is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria. The determination of the radiological response will be based on the investigator's reported evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy

REFERENCES:
- [Derived] Prete AA, Manca P, Messina M, Formica V, Frassineti GL, Zampino MG, Corsi DC, Orciuolo C, Prisciandaro M, Bergamo F, Angerilli V, Scartozzi M, Casagrande M, Masi G, Ronzoni M, Morano F, Vettore V, Salmaso R, Rasola C, Maddalena G, Del Bianco P, Milione M, Cremolini C, Fassan M, Pietrantonio F, Lonardi S. Extensive molecular profiling of squamous cell anal carcinoma in a phase 2 trial population: Translational analyses of the "CARACAS" study. Eur J Cancer. 2023 Mar;182:87-97. doi: 10.1016/j.ejca.2022.12.025. Epub 2023 Jan 9. PMID 36753836
- [Derived] Lonardi S, Prete AA, Morano F, Messina M, Formica V, Corsi DC, Orciuolo C, Frassineti GL, Zampino MG, Casagrande M, Masi G, Ronzoni M, Scartozzi M, Buonadonna A, Mosconi S, Ratti M, Sartore-Bianchi A, Tamburini E, Prisciandaro M, Bergamo F, Spada M, Corallo S, Vettore V, Loupakis F, Fassan M, Del Bianco P, Zagonel V, Pietrantonio F. Randomized phase II trial of avelumab alone or in combination with cetuximab for patients with previously treated, locally advanced, or metastatic squamous cell anal carcinoma: the CARACAS study. J Immunother Cancer. 2021 Nov;9(11):e002996. doi: 10.1136/jitc-2021-002996. PMID 34815354